CLINICAL TRIAL: NCT07382934
Title: Prevalence of Radix Entomolaris and Middle Mesial Canal in Lower Permanent Molars in an Egyptian Sub-Population Using CBCT: Cross Sectional Study
Brief Title: Prevalence of Radix Entomolaris and Middle Mesial Canal in an Egyptian Sub-population Using Cbct.
Acronym: RE MMC CBCT
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Ayman Ali, Postgraduate student, Cairo University
Other Study IDs: ENDO1-1-1
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Radix Entomolaris; Middle Mesial Canal
Keywords: the prevalence of RE and MMCs in mandibular first and second molars among an Egyptian sub- population.

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lower Permanent Molars in an Egyptian Sub- Population: Egyptian Sub- Population

SUMMARY:
The aim of the study is to determine the prevalence of RE and MMCs in mandibular first and second molars among an Egyptian sub- population.

DETAILED DESCRIPTION:
Primary Objective is to determine the prevalence of RE and MMC in mandibular molars within an Egyptian sub_population using CBCT analysis.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 years and above.
* Egyptian individuals with permanent mandibular molars had CBCT imaging.
* High-quality CBCT scans with clear visualization of mandibular molars.

Exclusion Criteria:

* Non- Egyptian patients.
* Molars are badly broken down with root defect such as root caries, or root resorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Egyptian sub-population
Sampling Method: Non-Probability Sample
Enrollment: 395 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Radix Entomolaris in Lower Permanent Molars | 1 year
  frequency and percentage of the prevalence of Radix Entomolaris

SECONDARY OUTCOMES:
Prevalence of Middle Mesial Canal in Lower Permanent Molars in an Egyptian Sub- Population Using CBCT: Cross Sectional Study. | 1 year
  Using CBCT to determine the prevalence of and Middle Mesial Canal frequency and prevalence in Lower Permanent Molars.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Talabani RM, Abdalrahman KO, Abdul RJ, Babarasul DO, Hilmi Kazzaz S. Evaluation of Radix Entomolaris and Middle Mesial Canal in Mandibular Permanent First Molars in an Iraqi Subpopulation Using Cone-Beam Computed Tomography. Biomed Res Int. 2022 Jul 11;2022:7825948. doi: 10.1155/2022/7825948. PMID: 35860794; PMCID: PMC9293536.